CLINICAL TRIAL: NCT00907569
Title: A Clinical Trial of Increased Chest Radiotherapy Dose for Limited Stage Small Cell Lung Cancer
Brief Title: Hypofractionated Radiotherapy for Limited Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24762
Record Dates: First submitted 2009-05-20; First posted 2009-05-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2011-09

CONDITIONS: Lung Neoplasm; Small Cell Carcinoma
Keywords: Small cell lung cancer; radiotherapy dose escalation
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Small Cell; Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: Hypofractionated Chest Radiotherapy — Hypofractionated chest radiotherapy regimen of 58 Gy delivered in 25 fractions in 5 weeks.

SUMMARY:
It is accepted that giving higher doses of chest radiation in as short a time span as possible improves chances of cure. In this study, the investigators propose to give an increased dose of chest radiotherapy for limited stage small cell lung cancer patients using a strategy of giving a slightly higher daily dose of radiotherapy than normal. The investigators hypothesize that our proposed chest radiotherapy dose will improve 2-year overall survival rates in patients with limited stage small cell lung cancer.

DETAILED DESCRIPTION:
The ideal chest radiotherapy dose/fractionation scheme for limited stage small cell lung cancer is undefined. Strategies of radiotherapy dose intensification with minimization of overall treatment time are felt to improve cure rates for LS-SCLC. Hypofractionation (giving higher than standard daily doses) facilitates both of these goals. In this study, we propose to use a dose escalated hypofractionated regimen of chest radiotherapy for patients with LS-SCLC.

ELIGIBILITY:
Inclusion Criteria:

* limited stage small cell lung cancer
* adequate pulmonary function test (FEV1 >1.0 L, DLCO >50%)
* signed study consent
* age at least 18 years
* Karnofsky performance status as least 70%
* eligible to receive standard concurrent small cell cancer chemotherapy

Exclusion Criteria:

* extensive stage disease
* mixed non small cell and small cell histology
* inadequate pulmonary function tests
* not eligible for concurrent chemotherapy
* subtotal or total tumor resection
* previous chest/neck radiotherapy
* prior or concurrent malignancy except non-melanomatous skin unless disease free for last 5 years
* pregnant
* prior chemotherapy for another malignancy
* patients with myocardial infarction within the preceding 6 months of symptomatic heart disease, including, angina, congestive heart failure, uncontrolled arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
2-year overall survival | 2011

SECONDARY OUTCOMES:
Quality of life | 2011
Patterns of Failure | 2011

CONTACTS AND LOCATIONS:
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada